CLINICAL TRIAL: NCT01245387
Title: Long-Term Non-Interventional Study (AB Study) To Investigate The Efficacy And Safety Of Macugen® In Patients With Neovascular Age-Related Macular Degeneration Under Conditions Of Routine Clinical Practice
Brief Title: Observational Study Of The Long-Term Effect Of Macugen In Patients With Wet Age-Related Macular Degeneration
Acronym: MACULA
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Other Study IDs: A5751021
Record Dates: First submitted 2010-09-29; First posted 2010-11-22 (Estimated); Results first posted 2011-01-07 (Estimated); Last update posted 2011-01-13 (Estimated); Status verified 2011-01

CONDITIONS: Macular Degeneration; Age-related Macular Degeneration; Neovascular Macular Degeneration
Keywords: prospective; observational; Phase 4; non-interventional; open-label
MeSH Terms: conditions — Macular Degeneration | interventions — pegaptanib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Macugen
  Interventions: Drug: Pegaptanib

INTERVENTIONS:
Drug: Pegaptanib — Dosage recommendations for MACUGEN took place on the basis of the approved Summary of Product Characteristics (SmPC) and were adjusted solely according to medical practice. MACUGEN® is available as pre-filled syringe containing 0.3 mg MACUGEN® in 90 µL injection solution for intravitreal injection. Macugen injections were documented to reflect the routine clinical practice. Follow-up visits were only carried out and documented if they took place as part of the standard medical treatment for the respective case and were necessary for medical and/or therapeutic reasons.

SUMMARY:
Long-term observational study to assess the safety, efficacy and quality of life of patients with neovascular age-related macular degeneration (AMD) under Macugen treatment.

DETAILED DESCRIPTION:
Ophthalmologists who are experienced in doing intravitreal injections in Germany

ELIGIBILITY:
Inclusion Criteria:

* patients with neovascular age-related macular degeneration

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with neovascular age-related macular degeneration
Sampling Method: Non-Probability Sample
Enrollment: 1001 (Actual)
Dates: Start 2006-08; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A5751021&StudyName=Observational%20Study%20Of%20The%20Long-Term%20Effect%20Of%20Macugen%20In%20Patients%20With%20Wet%20Age-Related%20Macular%20Degeneration%20

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This observational study did not define endpoints as primary or secondary. All endpoints arbitrarily assigned as primary for reporting results.
Groups:
- Macugen: Intraocular injections of Macugen (pegaptanib) into the study eye. The usage and dosage recommendations were in accordance with the Summary of Product Characteristics (SmPC) and based exclusively on the medical and therapeutic needs.
Period: Overall Study
Arm/Group | Macugen
Started | 1001
Completed | 188
Not Completed | 813
Not completed — Lost to Follow-up | 106
Not completed — Lack of Efficacy | 195
Not completed — Adverse Event | 9
Not completed — Death | 3
Not completed — Other | 131
Not completed — Missing discontinuation status | 369

BASELINE CHARACTERISTICS:
Arm/Group | Macugen
Number analyzed (Participants) | 1001
Age Continuous [Mean (Standard Deviation); unit: years] | 77.4 (7.8)
Sex/Gender, Customized [Number; unit: participants]
  Female | 666
  Male | 330
  Unspecified | 5

OUTCOME MEASURES:

1. Primary Outcome: Visual Acuity (VA)
Description: VA measured at each follow-up visit as the number of lines read on a standard eye chart (Snellen or Early Treatment Diabetic Retinopathy Study [EDTRS]) using a 5 meter distance, 1 meter distance, or verifying if participant was able to count fingers, perceive hand motion, or light. Follow-up visits occurred only if considered part of standard medical treatment. The timeframe was as follows: Visit 1: before first injection; Visit 2: first injection; Visit 3: 6 weeks after first injection (second injection).
Time Frame: Baseline, every 6 weeks up to Month 24 or early termination
Population: Full Analysis Set (FAS):participants who received at least 1 Macugen (pegaptanib) injection and had at least 1 VA measurement postbaseline. Participants with light perception or no light perception any time during study were excluded from FAS; N=participants with evaluable data; Last Visit: last available postbaseline value.
Measure: Mean (Standard Deviation); unit: lines of VA
Arm/Group | Macugen
Number analyzed (Participants) | 812
lines of VA
  Visit 1, Baseline (N=812) | 8.51 (5.03)
  Visit 2, Week 0, first injection (N=812) | 8.72 (5.19)
  Visit 3, Week 6 (N=785) | 8.67 (4.90)
  Visit 4, Week 12 (N=684) | 8.93 (4.97)
  Visit 5, Week 18 (N=537) | 9.06 (4.81)
  Visit 6, Week 24 (N=253) | 8.83 (5.32)
  Visit 7, Week 30 (N=203) | 8.60 (4.69)
  Visit 8, Week 36 (N=133) | 8.07 (3.81)
  Visit 9, Week 42 (N=86) | 8.35 (3.42)
  Visit 10, Week 48 (N=54) | 8.33 (3.44)
  Visit 11, Week 54 (N=11) | 8.86 (3.30)
  Visit 12, Week 60 (N=6) | 9.34 (3.33)
  Visit 13, Week 66 (N=4) | 8.49 (3.01)
  Visit 14, Week 72 (N=2) | 7.61 (3.37)
  Last Visit (N=786) | 9.26 (5.24)

2. Primary Outcome: Vision-related Functioning and Quality of Life Using the National Eye Institute Visual Functioning Questionnaire-25 (NEI-VFQ-25): Overall Composite Score
Description: Participant-reported vision-related functioning and quality of life measured using the 25 item NEI-VFQ-25. Converted scale 0-100 where higher score represented better functioning: General Health: item 1; General Vision: item 2; Ocular Pain: 4,19; Near Vision: 5,6,7; Distance Vision: 8,9,14; Social Functioning: 11,13; Mental Health Activities: 3,21,22,25; Role Difficulties: 17,18; Dependency: 20,23,24; Driving: 15c,16, 16a; Color Vision: 12; Peripheral Vision: 10.
Time Frame: Baseline, every 6 months up to Month 24 or early termination
Population: FAS; N=number of participants with evaluable data; Last Visit: last available postbaseline value.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Macugen
Number analyzed (Participants) | 485
Scores on a scale
  Visit 1, Baseline (N=485) | 54.05 (23.50)
  Visit 2, Month 6 (N=219) | 55.56 (22.17)
  Visit 3, Month 12 (N=167) | 57.13 (21.60)
  Visit 4, Month 18 (N=135) | 56.95 (20.58)
  Visit 5, Month 24 (N=338) | 56.09 (23.73)
  Last Visit (N=410) | 54.90 (23.86)

3. Primary Outcome: Number of Participants With Investigator Assessments of Efficacy
Description: Investigator's categorical assessment of the efficacy of Macugen (pegaptanib) treatment at the final visit or termination of therapy; Categories included Very Good, Good, Moderate, and Poor.
Time Frame: Month 24 or early termination
Population: FAS; N = number of participants with evaluable data.
Measure: Number; unit: Participants
Arm/Group | Macugen
Number analyzed (Participants) | 604
Participants
  Very Good | 36
  Good | 226
  Moderate | 168
  Poor | 174

4. Primary Outcome: Lesion Size (Number of Optic Disc Areas)
Description: Lesion size measured by Investigator after each injection as part of standard of care (SOC), using standard clinical methods practiced (fluorescein or indocyanine green angiography); Reported as the number of optic-disk areas, each of which were 2.54 millimeters squared (mm^2). Lesion size included choroidal neovascularization, exudation area, and hemorrhage, if present. The timeframe was as follows: Visit 1: before first injection; Visit 3: 6 weeks after first injection (second injection).
Time Frame: Baseline, every 6 weeks up to Month 24 or early termination
Population: FAS; N=number of participants with evaluable data; Last Visit: last available postbaseline value.
Measure: Mean (Standard Deviation); unit: number of optic disc areas
Arm/Group | Macugen
Number analyzed (Participants) | 712
number of optic disc areas
  Visit 1, Baseline (N=712) | 2.4 (1.6)
  Visit 3, Week 6 (N=190) | 2.1 (1.2)
  Visit 4, Week 12 (N=173) | 2.3 (1.7)
  Visit 5, Week 18 (N=316) | 2.2 (2.0)
  Visit 6, Week 24 (N=45) | 2.3 (1.3)
  Visit 7, Week 30 (N=45) | 3.2 (2.1)
  Visit 8, Week 36 (N=78) | 2.8 (2.0)
  Visit 9, Week 42 (N=15) | 2.5 (1.3)
  Visit 10, Week 48 (N=9) | 2.5 (1.4)
  Visit 11, Week 54 (N=6) | 2.3 (0.8)
  Visit 12, Week 60 (N=2) | 2.0 (1.4)
  Visit 13, Week 66 (N=3) | 0.8 (0.3)
  Last Visit (N=513) | 2.5 (2.1)

5. Primary Outcome: Number of Participants With a Change in Activity of Neovascular Membrane at Week 6
Description: Neovascular membrane activity (measured by leakage) assessed by Investigator at Visit 3, as part of SOC, using standard clinical methods practiced (fluorescein or indocyanine green angiography); Categories included increased, unchanged or decreased neovascular membrane activity.
Time Frame: Week 6
Population: FAS; N=number of participants with evaluable data.
Measure: Number; unit: Participants
Arm/Group | Macugen
Number analyzed (Participants) | 190
Participants
  Increased | 28
  Unchanged | 74
  Decreased | 88

6. Primary Outcome: Number of Participants With a Change in Activity of Neovascular Membrane at Week 12
Description: Neovascular membrane activity (measured by leakage) assessed by Investigator at Visit 4, as part of SOC, using standard clinical methods practiced (fluorescein or indocyanine green angiography); Categories included increased, unchanged or decreased neovascular membrane activity.
Time Frame: Week 12
Population: FAS; N=number of participants with evaluable data.
Measure: Number; unit: Participants
Arm/Group | Macugen
Number analyzed (Participants) | 173
Participants
  Increased | 22
  Unchanged | 66
  Decreased | 85

7. Primary Outcome: Number of Participants With a Change in Activity of Neovascular Membrane at Week 18
Description: Neovascular membrane activity (measured by leakage) assessed by Investigator at Visit 5, as part of SOC, using standard clinical methods practiced (fluorescein or indocyanine green angiography); Categories included increased, unchanged or decreased neovascular membrane activity.
Time Frame: Week 18
Population: FAS; N=number of participants with evaluable data.
Measure: Number; unit: Participants
Arm/Group | Macugen
Number analyzed (Participants) | 316
Participants
  Increased | 57
  Unchanged | 83
  Decreased | 176

8. Primary Outcome: Number of Participants With a Change in Activity of Neovascular Membrane at Week 24
Description: Neovascular membrane activity (measured by leakage) assessed by Investigator at Visit 6, as part of SOC, using standard clinical methods practiced (fluorescein or indocyanine green angiography); Categories included increased, unchanged or decreased neovascular membrane activity.
Time Frame: Week 24
Population: FAS; N=number of participants with evaluable data.
Measure: Number; unit: Participants
Arm/Group | Macugen
Number analyzed (Participants) | 46
Participants
  Increased | 13
  Unchanged | 15
  Decreased | 18

9. Primary Outcome: Number of Participants With a Change in Activity of Neovascular Membrane at Week 30
Description: Neovascular membrane activity (measured by leakage) assessed by Investigator at Visit 7, as part of SOC, using standard clinical methods practiced (fluorescein or indocyanine green angiography); Categories included increased, unchanged or decreased neovascular membrane activity.
Time Frame: Week 30
Population: FAS; N=number of participants with evaluable data.
Measure: Number; unit: Participants
Arm/Group | Macugen
Number analyzed (Participants) | 45
Participants
  Increased | 6
  Unchanged | 15
  Decreased | 24

10. Primary Outcome: Number of Participants With a Change in Activity of Neovascular Membrane at Week 36
Description: Neovascular membrane activity (measured by leakage) assessed by Investigator at Visit 8, as part of SOC, using standard clinical methods practiced (fluorescein or indocyanine green angiography); Categories included increased, unchanged or decreased neovascular membrane activity.
Time Frame: Week 36
Population: FAS; N=number of participants with evaluable data.
Measure: Number; unit: Participants
Arm/Group | Macugen
Number analyzed (Participants) | 78
Participants
  Increased | 11
  Unchanged | 21
  Decreased | 46

11. Primary Outcome: Number of Participants With a Change in Activity of Neovascular Membrane at Week 42
Description: Neovascular membrane activity (measured by leakage) assessed by Investigator at Visit 9, as part of SOC, using standard clinical methods practiced (fluorescein or indocyanine green angiography); Categories included increased, unchanged or decreased neovascular membrane activity.
Time Frame: Week 42
Population: FAS; N=number of participants with evaluable data.
Measure: Number; unit: Participants
Arm/Group | Macugen
Number analyzed (Participants) | 15
Participants
  Increased | 3
  Unchanged | 6
  Decreased | 6

12. Primary Outcome: Number of Participants With a Change in Activity of Neovascular Membrane at Week 48
Description: Neovascular membrane activity (measured by leakage) assessed by Investigator at Visit 10, as part of SOC, using standard clinical methods practiced (fluorescein or indocyanine green angiography); Categories included increased, unchanged or decreased neovascular membrane activity.
Time Frame: Week 48
Population: FAS; N=number of participants with evaluable data.
Measure: Number; unit: Participants
Arm/Group | Macugen
Number analyzed (Participants) | 10
Participants
  Increased | 2
  Unchanged | 3
  Decreased | 5

13. Primary Outcome: Number of Participants With a Change in Activity of Neovascular Membrane at Week 54
Description: Neovascular membrane activity (measured by leakage) assessed by Investigator at Visit 11, as part of SOC, using standard clinical methods practiced (fluorescein or indocyanine green angiography); Categories included increased, unchanged or decreased neovascular membrane activity.
Time Frame: Week 54
Population: FAS; N=number of participants with evaluable data.
Measure: Number; unit: Participants
Arm/Group | Macugen
Number analyzed (Participants) | 6
Participants
  Increased | 0
  Unchanged | 2
  Decreased | 4

14. Primary Outcome: Number of Participants With a Change in Activity of Neovascular Membrane at Week 60
Description: Neovascular membrane activity (measured by leakage) assessed by Investigator at Visit 12, as part of SOC, using standard clinical methods practiced (fluorescein or indocyanine green angiography); Categories included increased, unchanged or decreased neovascular membrane activity.
Time Frame: Week 60
Population: FAS; N=number of participants with evaluable data.
Measure: Number; unit: Participants
Arm/Group | Macugen
Number analyzed (Participants) | 2
Participants
  Increased | 1
  Unchanged | 0
  Decreased | 1

15. Primary Outcome: Number of Participants With a Change in Activity of Neovascular Membrane at Week 66
Description: Neovascular membrane activity (measured by leakage) assessed by Investigator at Visit 13, as part of SOC, using standard clinical methods practiced (fluorescein or indocyanine green angiography); Categories included increased, unchanged or decreased neovascular membrane activity.
Time Frame: Week 66
Population: FAS; N=number of participants with evaluable data.
Measure: Number; unit: Participants
Arm/Group | Macugen
Number analyzed (Participants) | 3
Participants
  Increased | 0
  Unchanged | 1
  Decreased | 2

16. Primary Outcome: Number of Participants With a Change in Activity of Neovascular Membrane at Week 72
Description: Neovascular membrane activity (measured by leakage) assessed by Investigator at Visit 14, as part of SOC, using standard clinical methods practiced (fluorescein or indocyanine green angiography); Categories included increased, unchanged or decreased neovascular membrane activity.
Time Frame: Week 72
Population: FAS; N=number of participants with evaluable data.
Measure: Number; unit: Participants
Arm/Group | Macugen
Number analyzed (Participants) | 1
Participants
  Increased | 0
  Unchanged | 0
  Decreased | 1

17. Primary Outcome: Number of Participants With a Change in Activity of Neovascular Membrane at Last Visit
Description: Neovascular membrane activity (measured by leakage) assessed by Investigator at the Last Visit, as part of SOC, using standard clinical methods practiced (fluorescein or indocyanine green angiography); Categories included increased, unchanged or decreased neovascular membrane activity. Last Visit: last available postbaseline value.
Time Frame: Month 24 or early termination
Population: FAS; N=number of participants with evaluable data.
Measure: Number; unit: Participants
Arm/Group | Macugen
Number analyzed (Participants) | 514
Participants
  Increased | 101
  Unchanged | 170
  Decreased | 243

18. Primary Outcome: Number of Participants With Pigment Epithelial Detachment (PED) at Baseline
Description: PED assessed by Investigator at baseline as part of SOC for participants with age-related macular degeneration; Standard clinical methods practiced (fluorescein or indocyanine green angiography); Categories included present or absent.
Time Frame: Baseline
Population: FAS; N=number of participants with evaluable data.
Measure: Number; unit: Participants
Arm/Group | Macugen
Number analyzed (Participants) | 713
Participants
  Present | 240
  Absent | 473

19. Primary Outcome: Number of Participants With PED at Week 6
Description: PED assessed by Investigator at Visit 3, as part of SOC, using standard clinical methods practiced (fluorescein or indocyanine green angiography); Categories included present or absent.
Time Frame: Week 6
Population: FAS; N=number of participants with evaluable data.
Measure: Number; unit: Participants
Arm/Group | Macugen
Number analyzed (Participants) | 188
Participants
  Present | 46
  Absent | 142

20. Primary Outcome: Number of Participants With PED at Week 12
Description: PED assessed by Investigator at Visit 4, as part of SOC, using standard clinical methods practiced (fluorescein or indocyanine green angiography); Categories included present or absent.
Time Frame: Week 12
Population: FAS; N=number of participants with evaluable data.
Measure: Number; unit: Participants
Arm/Group | Macugen
Number analyzed (Participants) | 169
Participants
  Present | 32
  Absent | 137

21. Primary Outcome: Number of Participants With PED at Week 18
Description: PED assessed by Investigator at Visit 5, as part of SOC, using standard clinical methods practiced (fluorescein or indocyanine green angiography); Categories included present or absent.
Time Frame: Week 18
Population: FAS; N=number of participants with evaluable data.
Measure: Number; unit: Participants
Arm/Group | Macugen
Number analyzed (Participants) | 313
Participants
  Present | 45
  Absent | 268

22. Primary Outcome: Number of Participants With PED at Week 24
Description: PED assessed by Investigator at Visit 6, as part of SOC, using standard clinical methods practiced (fluorescein or indocyanine green angiography); Categories included present or absent.
Time Frame: Week 24
Population: FAS; N=number of participants with evaluable data.
Measure: Number; unit: Participants
Arm/Group | Macugen
Number analyzed (Participants) | 45
Participants
  Present | 7
  Absent | 38

23. Primary Outcome: Number of Participants With PED at Week 30
Description: PED assessed by Investigator at Visit 7, as part of SOC, using standard clinical methods practiced (fluorescein or indocyanine green angiography); Categories included present or absent.
Time Frame: Week 30
Population: FAS; N=number of participants with evaluable data.
Measure: Number; unit: Participants
Arm/Group | Macugen
Number analyzed (Participants) | 44
Participants
  Present | 11
  Absent | 33

24. Primary Outcome: Number of Participants With PED at Week 36
Description: PED assessed by Investigator at Visit 8, as part of SOC, using standard clinical methods practiced (fluorescein or indocyanine green angiography); Categories included present or absent.
Time Frame: Week 36
Population: FAS; N=number of participants with evaluable data.
Measure: Number; unit: Participants
Arm/Group | Macugen
Number analyzed (Participants) | 77
Participants
  Present | 11
  Absent | 66

25. Primary Outcome: Number of Participants With PED at Week 42
Description: PED assessed by Investigator at Visit 9, as part of SOC, using standard clinical methods practiced (fluorescein or indocyanine green angiography); Categories included present or absent.
Time Frame: Week 42
Population: FAS; N=number of participants with evaluable data.
Measure: Number; unit: Participants
Arm/Group | Macugen
Number analyzed (Participants) | 15
Participants
  Present | 3
  Absent | 12

26. Primary Outcome: Number of Participants With PED at Week 48
Description: PED assessed by Investigator at Visit 10, as part of SOC, using standard clinical methods practiced (fluorescein or indocyanine green angiography); Categories included present or absent.
Time Frame: Week 48
Population: FAS; N=number of participants with evaluable data.
Measure: Number; unit: Participants
Arm/Group | Macugen
Number analyzed (Participants) | 10
Participants
  Present | 6
  Absent | 4

27. Primary Outcome: Number of Participants With PED at Week 54
Description: PED assessed by Investigator Visit 11, as part of SOC, using standard clinical methods practiced (fluorescein or indocyanine green angiography); Categories included present or absent.
Time Frame: Week 54
Population: FAS; N=number of participants with evaluable data.
Measure: Number; unit: Participants
Arm/Group | Macugen
Number analyzed (Participants) | 6
Participants
  Present | 1
  Absent | 5

28. Primary Outcome: Number of Participants With PED at Last Visit
Description: PED assessed by Investigator at Last Visit, as part of SOC, using standard clinical methods practiced (fluorescein or indocyanine green angiography); Categories included present or absent. Last Visit: last available postbaseline value.
Time Frame: Month 24 or early termination
Population: FAS; N=number of participants with evaluable data.
Measure: Number; unit: Participants
Arm/Group | Macugen
Number analyzed (Participants) | 509
Participants
  Present | 87
  Absent | 422

29. Primary Outcome: Central Retinal Thickness
Description: Central retinal thickness assessed by Investigator every 6 weeks, as part of SOC, using standard clinical methods practiced (optical coherence tomography) and reported as mean central retinal thickness. The timeframe was as follows: Visit 1: before first injection; Visit 3: 6 weeks after first injection (second injection).
Time Frame: Baseline, every 6 weeks up to Month 24 or early termination
Population: FAS; N=number of participants with evaluable data; Last Visit: last available postbaseline value.
Measure: Mean (Standard Deviation); unit: Micrometers (Mcm)
Arm/Group | Macugen
Number analyzed (Participants) | 316
Micrometers (Mcm)
  Visit 1, Baseline (N=316) | 309.2 (105.9)
  Visit 3, Week 6 (N=224) | 305.8 (111.3)
  Visit 4, Week 12 (N=173) | 307.3 (122.9)
  Visit 5, Week 18 (N=205) | 297.8 (145.0)
  Visit 6, Week 24 (N=33) | 328.9 (180.5)
  Visit 7, Week 30 (N=26) | 272.7 (67.4)
  Visit 8, Week 36 (N=27) | 319.6 (118.7)
  Visit 9, Week 42 (N=13) | 252.9 (88.8)
  Visit 10, Week 48 (N=3) | 312.0 (133.5)
  Last Visit (N=311) | 295.2 (138.5)

30. Primary Outcome: Number of Participants With Angiographic Subtype Reported at Baseline
Description: Angiographic subtype assessed by Investigator at Baseline, as part of SOC, using standard clinical methods practiced (fluorescein angiography or indocyanine green angiography) and the percent [%] classic fraction categories included unclear, occult (0% classic), minimally classic (1-49% classic), predominantly classic (50-99% classic), and pure classic (100% classic).
Time Frame: Baseline
Population: FAS; N=number of participants with evaluable data.
Measure: Number; unit: Participants
Arm/Group | Macugen
Number analyzed (Participants) | 716
Participants
  unclear | 76
  occult | 363
  minimally classic | 113
  predominantly classic | 138
  pure classic | 26

31. Primary Outcome: Number of Participants With Angiographic Subtype Reported at Week 6
Description: Angiographic subtype assessed by Investigator at Visit 3, as part of SOC, using standard clinical methods practiced (fluorescein angiography or indocyanine green angiography) and the percent [%] classic fraction categories included unclear, occult (0% classic), minimally classic (1-49% classic), predominantly classic (50-99% classic), and pure classic (100% classic).
Time Frame: Week 6
Population: FAS;N=number of participants with evaluable data.
Measure: Number; unit: Participants
Arm/Group | Macugen
Number analyzed (Participants) | 190
Participants
  unclear | 29
  occult | 81
  minimally classic | 21
  predominantly classic | 56
  pure classic | 3

32. Primary Outcome: Number of Participants With Angiographic Subtype Reported at Week 12
Description: Angiographic subtype assessed by Investigator at Visit 4, as part of SOC, using standard clinical methods practiced (fluorescein angiography or indocyanine green angiography) and the percent [%] classic fraction categories included unclear, occult (0% classic), minimally classic (1-49% classic), predominantly classic (50-99% classic), and pure classic (100% classic).
Time Frame: Week 12
Population: FAS; N=number of participants with evaluable data.
Measure: Number; unit: Participants
Arm/Group | Macugen
Number analyzed (Participants) | 173
Participants
  unclear | 29
  occult | 71
  minimally classic | 21
  predominantly classic | 50
  pure classic | 2

33. Primary Outcome: Number of Participants With Angiographic Subtype Reported at Week 18
Description: Angiographic subtype assessed by Investigator at Visit 5, as part of SOC, using standard clinical methods practiced (fluorescein angiography or indocyanine green angiography) and the percent [%] classic fraction categories included unclear, occult (0% classic), minimally classic (1-49% classic), predominantly classic (50-99% classic), and pure classic (100% classic).
Time Frame: Week 18
Population: FAS; N=number of participants with evaluable data.
Measure: Number; unit: Participants
Arm/Group | Macugen
Number analyzed (Participants) | 316
Participants
  unclear | 68
  occult | 140
  minimally classic | 70
  predominantly classic | 30
  pure classic | 8

34. Primary Outcome: Number of Participants With Angiographic Subtype Reported at Week 24
Description: Angiographic subtype assessed by Investigator at Visit 6, as part of SOC, using standard clinical methods practiced (fluorescein angiography or indocyanine green angiography) and the percent [%] classic fraction categories included unclear, occult (0% classic), minimally classic (1-49% classic), predominantly classic (50-99% classic), and pure classic (100% classic).
Time Frame: Week 24
Population: FAS; N=number of participants with evaluable data.
Measure: Number; unit: Participants
Arm/Group | Macugen
Number analyzed (Participants) | 45
Participants
  unclear | 7
  occult | 26
  minimally classic | 5
  predominantly classic | 5
  pure classic | 2

35. Primary Outcome: Number of Participants With Angiographic Subtype Reported at Week 30
Description: Angiographic subtype assessed by Investigator at Visit 7, as part of SOC, using standard clinical methods practiced (fluorescein angiography or indocyanine green angiography) and the percent (%) classic fraction categories included unclear, occult (0% classic), minimally classic (1-49% classic), predominantly classic (50-99% classic), and pure classic (100% classic).
Time Frame: Week 30
Population: FAS; N=number of participants with evaluable data.
Measure: Number; unit: Participants
Arm/Group | Macugen
Number analyzed (Participants) | 45
Participants
  unclear | 10
  occult | 23
  minimally classic | 8
  predominantly classic | 3
  pure classic | 1

36. Primary Outcome: Number of Participants With Angiographic Subtype Reported at Week 36
Description: Angiographic subtype assessed by Investigator at Visit 8, as part of SOC, using standard clinical methods practiced (fluorescein angiography or indocyanine green angiography) and the % classic fraction categories included unclear, occult (0% classic), minimally classic (1-49% classic), predominantly classic (50-99% classic), and pure classic (100% classic).
Time Frame: Week 36
Population: FAS; N=number of participants with evaluable data.
Measure: Number; unit: Participants
Arm/Group | Macugen
Number analyzed (Participants) | 78
Participants
  unclear | 5
  occult | 37
  minimally classic | 30
  predominantly classic | 3
  pure classic | 3

37. Primary Outcome: Number of Participants With Angiographic Subtype Reported at Week 42
Description: Angiographic subtype assessed by Investigator at Visit 9, as part of SOC, using standard clinical methods practiced (fluorescein angiography or indocyanine green angiography) and the % classic fraction categories included unclear, occult (0% classic), minimally classic (1-49% classic), predominantly classic (50-99% classic), and pure classic (100% classic).
Time Frame: Week 42
Population: FAS; N=number of participants with evaluable data.
Measure: Number; unit: Participants
Arm/Group | Macugen
Number analyzed (Participants) | 15
Participants
  unclear | 3
  occult | 10
  minimally classic | 1
  predominantly classic | 0
  pure classic | 1

38. Primary Outcome: Number of Participants With Angiographic Subtype Reported at Week 48
Description: Angiographic subtype assessed by Investigator at Visit 10, as part of SOC, using standard clinical methods practiced (fluorescein angiography or indocyanine green angiography) and the % classic fraction categories included unclear, occult (0% classic), minimally classic (1-49% classic), predominantly classic (50-99% classic), and pure classic (100% classic).
Time Frame: Week 48
Population: FAS; N=number of participants with evaluable data.
Measure: Number; unit: Participants
Arm/Group | Macugen
Number analyzed (Participants) | 10
Participants
  unclear | 0
  occult | 7
  minimally classic | 3
  predominantly classic | 0
  pure classic | 0

39. Primary Outcome: Number of Participants With Angiographic Subtype Reported at Week 54
Description: Angiographic subtype assessed by Investigator at Visit 11, as part of SOC, using standard clinical methods practiced (fluorescein angiography or indocyanine green angiography) and the % classic fraction categories included unclear, occult (0% classic), minimally classic (1-49% classic), predominantly classic (50-99% classic), and pure classic (100% classic).
Time Frame: Week 54
Population: FAS; N=number of participants with evaluable data.
Measure: Number; unit: Participants
Arm/Group | Macugen
Number analyzed (Participants) | 6
Participants
  unclear | 0
  occult | 3
  minimally classic | 3
  predominantly classic | 0
  pure classic | 0

40. Primary Outcome: Number of Participants With Angiographic Subtype Reported at Last Visit
Description: Angiographic subtype assessed by Investigator at the Last Visit, as part of SOC, using standard clinical methods practiced (fluorescein angiography or indocyanine green angiography) and the % classic fraction categories included unclear, occult (0% classic), minimally classic (1-49% classic), predominantly classic (50-99% classic), and pure classic (100% classic). Last Visit: last available postbaseline value.
Time Frame: Month 24 or early termination
Population: FAS; N=number of participants with evaluable data.
Measure: Number; unit: Participants
Arm/Group | Macugen
Number analyzed (Participants) | 514
Participants
  unclear | 105
  occult | 251
  minimally classic | 88
  predominantly classic | 58
  pure classic | 12

41. Other Pre Specified Outcome: Time to First Adverse Event (AE)
Description: Time to first AE during the study evaluated by Kaplan-Meier Product-limit methods. AE:any untoward medical occurrence in a participant administered a product or medical device in the context of study; the event need not necessarily have a causal relationship with the treatment or usage.
Time Frame: Baseline up to Month 24 or early termination
Population: Safety Set: all participants who received at least 1 Macugen (pegaptanib) injection and provided data post baseline. Data not analyzed due to low number of AEs.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Macugen
Number analyzed (Participants) | 0

42. Other Pre Specified Outcome: Number of Participants With Complications Associated With Injection
Description: Complications associated with injection during the study with onset at or after date of first injection was recorded by the Investigator.
Time Frame: Baseline up to Month 24 or early termination
Population: Safety Set; N=number of participants with evaluable data.
Measure: Number; unit: Participants
Arm/Group | Macugen
Number analyzed (Participants) | 815
Participants
  Yes | 1
  No | 814

43. Other Pre Specified Outcome: Treatment Tolerability
Description: Investigator's overall evaluation of tolerability; Categories included: Very Good, Good, Moderate, and Poor.
Time Frame: Month 24 or early termination
Population: Safety Set; N=number of participants with evaluable data.
Measure: Number; unit: Participants
Arm/Group | Macugen
Number analyzed (Participants) | 589
Participants
  Very Good | 182
  Good | 367
  Moderate | 35
  Poor | 5

44. Other Pre Specified Outcome: Intraocular Pressure (IOP)
Description: IOP measured at each visit using either applanation tonometry or non-contact before intraviterial injection, reported as pre-dose pressure of treated eye in millimeters of mercury (mmHg). The timeframe was as follows: Visit 1: IOP before any injection; Visit 2: IOP before first injection; Visit 3: IOP before second injection.
Time Frame: Baseline, every 6 weeks up to Month 24 or early termination
Population: Safety Set; N=number of participants with evaluable data; Last Visit: last available postbaseline value.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Macugen
Number analyzed (Participants) | 809
mmHg
  Visit 1, Baseline (N=809) | 15.7 (2.8)
  Visit 2, Week 0 (N=568) | 15.7 (3.0)
  Visit 3, Week 6 (N=772) | 15.7 (3.2)
  Visit 4, Week 12 (N=661) | 15.8 (3.1)
  Visit 5, Week 18 (N=505) | 15.9 (3.1)
  Visit 6, Week 24 (N=237) | 15.5 (2.8)
  Visit 7, Week 30 (N=190) | 15.5 (2.6)
  Visit 8, Week 36 (N=123) | 15.8 (2.3)
  Visit 9, Week 42 (N=80) | 15.4 (2.0)
  Visit 10, Week 48 (N=53) | 15.7 (2.3)
  Visit 11, Week 54 (N=11) | 16.3 (2.9)
  Visit 12, Week 60 (N=6) | 15.3 (4.0)
  Visit 13, Week 66 (N=4) | 18.0 (2.3)
  Visit 14, Week 72 (N=2) | 17.0 (1.4)
  Last Visit (N=776) | 15.6 (3.0)

45. Other Pre Specified Outcome: Change in IOP Between Predose and Postdose Assessment
Description: IOP measured at each visit using either applanation tonometry or non-contact before and after intraviterial injection. Change in IOP equals postdose IOP minus predose IOP.
Time Frame: Baseline, every 6 weeks up to Month 24 or early termination
Population: Safety Set; N=number of participants with evaluable data; Last Visit: last available postbaseline value.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Macugen
Number analyzed (Participants) | 718
mmHg
  Visit 2, Week 0 (N=559) | 1.3 (3.7)
  Visit 3, Week 6 (N=704) | 1.3 (4.1)
  Visit 4, Week 12 (N=600) | 1.3 (3.8)
  Visit 5, Week 18 (N=240) | 1.4 (3.7)
  Visit 6, Week 24 (N=210) | 1.5 (3.3)
  Visit 7, Week 30 (N=158) | 2.4 (4.9)
  Visit 8, Week 36 (N=90) | 1.8 (2.5)
  Visit 9, Week 42 (N=63) | 2.2 (2.8)
  Visit 10, Week 48 (N=48) | 2.3 (2.1)
  Visit 11, Week 54 (n=7) | 1.3 (1.7)
  Visit 12, Week 60 (N=4) | 1.3 (6.3)
  Visit 13, Week 66 (N=2) | -2.0 (4.2)
  Last Visit (N=718) | 1.4 (3.9)

46. Other Pre Specified Outcome: IOP Mean Difference (Within a Participant)
Description: Average predose minus postdose mean difference in IOP within a participant
Time Frame: Baseline, every 6 weeks up to Month 24 or early termination
Population: Safety Set; N=number of participants with evaluable data.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Macugen
Number analyzed (Participants) | 763
mmHg | 1.3 (2.9)

ADVERSE EVENTS:
Description: The Safety population (N=816) is less than total number of participants in study (1001) because some participants had a baseline visit but no injection or no data post baseline. The same event may appear as both an adverse event (AE) and a serious adverse event (SAE). However, what is presented are distinct events.
Arm/Group | Macugen
Serious Adverse Events (participants affected / at risk) | 16/816
Other Adverse Events (participants affected / at risk) | 12/816
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Macugen (N=816)
Endophthalmitis (Infections and infestations) | 4
Sepsis (Infections and infestations) | 1
Myocardial infarction (Cardiac disorders) | 2
Atrial fibrillation (Cardiac disorders) | 1
Cardiac failure (Cardiac disorders) | 1
Coronary artery disease (Cardiac disorders) | 1
Retinal haemorrhage (Eye disorders) | 3
Choroidal neovascularisation (Eye disorders) | 1
Retinal detachment (Eye disorders) | 1
Retinal tear (Eye disorders) | 1
Cerebrovascular accident (Nervous system disorders) | 3
Nausea (Gastrointestinal disorders) | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Macugen (N=816)
Visual acuity reduced (Eye disorders) | 6
Retinal haemorrhage (Eye disorders) | 1
Choroidal neovascularisation (Eye disorders) | 1
Retinal detachment (Eye disorders) | 1
Detachment of retinal pigment epithelium (Eye disorders) | 1
Glaucoma (Eye disorders) | 1
Subretinal fibrosis (Eye disorders) | 1
Vitreous haemorrhage (Eye disorders) | 1
Endophthalmitis (Infections and infestations) | 1
Intraocular pressure increased (Investigations) | 2
Paracentesis eye (Investigations) | 1
Injection site reaction (General disorders) | 1
Eye operation (Surgical and medical procedures) | 1

LIMITATIONS AND CAVEATS:
Time to first AE not estimated due to insufficient number of events. Visit numbers for NEI-VFQ-25 deviated from numbering used in other analyses; it represents the sequence number of questionaries administered (Visit 1=first assessment, etc.).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.